CLINICAL TRIAL: NCT03220542
Title: The Effect of Broccoli Sprout Extract and Probiotics on Proton Pump Inhibitor-based Triple Therapy for Eradication of Helicobacter Pylori: a Prospective Randomized Trial
Brief Title: The Effect of Broccoli Sprout Extract and Probiotics for Eradication of Helicobacter Pylori
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Jung-Wook Kim, Clinical assistant professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Broccoli2014
Record Dates: First submitted 2017-07-09; First posted 2017-07-18 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter Pylori; Probiotics; Sulforaphane
MeSH Terms: interventions — Probiotics; sulforaphane; Esomeprazole; Amoxicillin; Clarithromycin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Probiotics (Experimental): Saccharomyces boulardii + Esomeprazole + Amoxicillin + Clarithromycin
  Interventions: Drug: Probiotics; Drug: Esomeprazole; Drug: Amoxicillin; Drug: Clarithromycin
- Broccoli (Experimental): Broccoli Sprouts Extract + Esomeprazole + Amoxicillin + Clarithromycin
  Interventions: Dietary Supplement: Broccoli; Drug: Esomeprazole; Drug: Amoxicillin; Drug: Clarithromycin
- Triple Therapy (Active Comparator): Esomeprazole + Amoxicillin + Clarithromycin
  Interventions: Drug: Esomeprazole; Drug: Amoxicillin; Drug: Clarithromycin

INTERVENTIONS:
Drug: Probiotics — Saccharomyces boulardii
  Other Names: Bioflor 250, Kuhnil Pharmacy, Seoul, Korea
  Arms: Probiotics
Dietary Supplement: Broccoli — Broccoli sprouts extract
  Other Names: Sulforaphane
  Arms: Broccoli
Drug: Esomeprazole — Esomeprazole
Drug: Amoxicillin — Amoxicillin
Drug: Clarithromycin — Clarithromycin

SUMMARY:
In Korea, the first-line therapy to treat Helicobacter pylori (Hp) consists of a proton pump inhibitor (PPI) and two antibiotics for one week. But, eradication has become less successful due to low compliance and high resistance to the antibiotics. Therefore, it is necessary to develop new treatment strategies that increase the eradication rate and reduce adverse effects. In vitro study, we previously reported that a broccoli sprout extract containing sulforaphane may prevent lipid peroxidation in the gastric mucosa and play a cytoprotective role in Hp-induced gastritis. Also, several studies suggested that probiotics could be effective for improving Hp eradication rate or reducing adverse events. But, their effect for eradication of Hp is not yet conclusive. The aims of this prospective study is to investigate the efficacy of a broccoli sprout extract containing sulforaphane and probiotics for eradication of Hp, compared with standard triple therapy.

ELIGIBILITY:
Inclusion Criteria:

* Helicobacter pylori infected patients
* Patients with active or healing gastric/duodenal ulcers

Exclusion Criteria:

* prior Hp eradication therapy
* previous gastric resection
* previous use of proton pump inhibitors, bismuth, H2 receptor antagonist or antibiotics within 4 weeks of the study
* Patients who were pregnant or lactating

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori eradication | 5 weeks after treatment initiation
  Using the urea breath test

CONTACTS AND LOCATIONS:
Locations (1):
- Kyung Hee University Hospital, Seoul, South Korea